CLINICAL TRIAL: NCT04209959
Title: Comparison of Efficacy and Safety of Different Doses of Nifekalant Instant Cardioversion of Persistent Atrial Fibrillation During Radiofrequency Ablation：a Single-center Randomized Controlled Trial
Brief Title: Comparison of Efficacy and Safety of Different Doses of Nifekalant Instant Cardioversion of Persistent Atrial Fibrillation During Radiofrequency Ablation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014[023]
Record Dates: First submitted 2019-12-03; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — nifekalant

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low dose group (Experimental)
  Interventions: Drug: nifekalant
- middle dose group (Experimental)
  Interventions: Drug: nifekalant
- high dose group (Experimental)
  Interventions: Drug: nifekalant

INTERVENTIONS:
Drug: nifekalant — Nifekalant was randomly given intravenously as a loading dose of 0.3 mg/kg, 0.4 mg/kg, or 0.5 mg/kg for five minutes without the continuous infusion for all study population, while blood pressure, surface electrocardiograms (ECG), intracardiac electrograms were monitored for half an hour. While nifekalant was given intravenously, QT interval, QTc interval and RR interval were recorded at 0, 1, 3, 5, 10, 15, 20 and 30minutes, respectively, because drug action almost disappeared within 30minutes since a single dose of intravenous nifekalant injection. These doses of nifekalant were determined based on the results of the previous study and the medicine operation instruction. Once AF continued after administration or Torsade de points was observed, external electrical cardioversion was given immediately.

SUMMARY:
Atrial fibrillation (AF) is one of the most common tachyarrhythmias with substantial morbidity, disability and mortality. It is estimated that the number of patients with AF is expected to reach 7 million by 2050. Radiofrequency catheter ablation (RFCA) are the effective treatment for patients with drug-refractory symptomatic paroxysmal or persistent AF. However, the successful rate of RFCA for persistent AF during the first procedure still relatively low, the investigators also need pharmacological cardioversion or external electrical conversion. Several studies showed intravenous nifekalant injection after RFCA provided relative high rate of sinus conversion during catheter ablation in paroxysmal or persistent AF. Nevertheless, there is still no acceptable universal opinion on which dosage of nifekalant is preferable for converting AF during the operation. In order to address this issue, the investigators initiated the study to evaluate the efficacy and safety of different doses of intravenous nifekalant injection in the rapid cardioversion of persistent AF during radiofrequency catheter ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common tachyarrhythmias with substantial morbidity, disability and mortality. Its prevalence increases with advanced age. About one percent of patients suffering from AF are younger than sixty years, twelve percent are between seventy-five and eighty-five years, and about thirty-three percent are older than eighty years. It is estimated that the number of patients with AF is expected to reach 7 million by 2050. At present, the medical anti-arrhythmic therapy and radiofrequency ablation have been as important treatment for patients with AF. Compared with the treatment of anti-arrhythmia therapy, radiofrequency ablation could significantly improve the rate of long-term AF-free survival. Thus, radiofrequency ablation has become the radical method for patients suffering AF.

However, the successful rate of first radiofrequency ablation for patients with persistent AF was only about 65%. Due to low sinus maintenance rate after catheter ablation, anti-arrhythmic drugs (AADs) or external electric cardioversion was used to converting atrial fibrillation during the procedure. Compared with traditional AADs for pharmacologic cardioversion, such as quinidine, propafenone and amiodarone, nifekalant is a new class III AADs for rapid cardioversion of persistent AF during radiofrequency ablation, and its prevalence of AF termination during procedure was approximately 64.6%. Nevertheless, the efficacy and safety of different doses of intravenous nifekalant injection in the rapid cardioversion of persistent AF during radiofrequency catheter ablation has not been tested in large, randomized, controlled trials, and guidelines provide no clear consensus regarding the best dose recommended.

In order to address this issue, the investigators initiated the study to evaluate the efficacy and safety of different doses of intravenous nifekalant injection in the rapid cardioversion of persistent AF during radiofrequency catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic persistent or longstanding persistent AF
* An absence of response to, unacceptable side effects from, or unwillingness to take antiarrhythmic agents
* Willingness to receive combined ablation strategy, including bilateral circumferential pulmonary vein isolation and linear ablation
* Failure to terminate AF to after combined ablation strategy
* Willingness to receive intravenous treatment with nifekalant during the procedure

Exclusion Criteria:

* A history of nontraumatic intracerebral hemorrhage at any time
* Gastrointestinal bleeding within the past six months
* Major surgery within thirty days
* A known bleeding diathesis or coagulation disorder
* A confirmed thrombus in the left atrium by esophageal ultrasound
* Renal failure requiring dialysis
* Pregnant or lactating
* A left ventricular ejection fraction (LVEF) of 30% or less
* Ventricular tachycardia with prolonged QT interval
* Patients with QTc interval of more than 500 ms
* Torsades de pointes (Tdp), or Brugada syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the successful rates of different doses of nifekalant instant cardioversion of persistent atrial fibrillation after radiofrequency ablation | up to 12 months
  Participants are randomized to one of three groups: low dose group (0.3mg/kg), middle dose group (0.4mg/kg), or high dose group (0.5mg/kg). The successful rates of different doses of nifekalant instant cardioversion were reported in terms of count and percentage, respectively.
The occurrence of adverse events, including sinus bradycardia, cardiac arrest, Torsade de points and ventricular fibrillation confirmed in standard 12-lead ECGs and intracardiac electrograms within 30 minutes among different treatment groups. | up to 12 months
  The occurrence of adverse events, such as sinus bradycardia, cardiac arrest, Torsade de points and ventricular fibrillation confirmed in standard 12-lead ECGs were represented in terms of count and percentage, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No